CLINICAL TRIAL: NCT01420198
Title: A Middle Eastern Immigrant Population At-risk for Diabetes; Contributing Risk Factors and the Efficiency and Cost-effectiveness of a Culturally Adopted Lifestyle Intervention Program - the MEDIM Study.
Brief Title: Efficiency and Cost-effectiveness of a Culturally Adopted Lifestyle Intervention Program - the MEDIM Study.
Acronym: MEDIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009/36
Record Dates: First submitted 2011-06-27; First posted 2011-08-19 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Type 2 Diabetes; Impaired Glucose Tolerance; Obesity; Physical Activity
Keywords: Diabetes type 2; Lifestyle intervention; QALY; Ethnic group; Impaired glucose tolerance; Impaired fasting glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle intervention (Experimental): Lifestyle intervention: 500 participants from Iraq with obesity and/or prediabetes (impaired fasting glucose) and we expect to recruit 308 participants. Half of them will be randomized to lifestyle intervention i.e. group counseling and physical activity during a period of 1 year. An equal amount of controls will have treatment as usual. Every third month blood tests and a physical exam will be conducted in the intervention group.
  Interventions: Behavioral: Lifestyle intervention
- Controls (No Intervention): Controls have treatment as usual. Every third month blood tests and a physical exam will be conducted in the control group.

INTERVENTIONS:
Behavioral: Lifestyle intervention — Increased physical activity and improved food habits
  Arms: Lifestyle intervention

SUMMARY:
An increasing proportion of Sweden's population comprises non-European immigrants, who constitute a high risk-population for T2D. Numbering almost 9,000 individuals, Iraqi citizens represent the largest immigrant group in Malmoe and are identified as a risk group for Type 2 Diabetes (T2D) in whom genetic and lifestyle factors probably play significant roles in the development of T2D.

Several studies have shown that adoption of an active lifestyle by at-risk individuals dramatically reduces the risk of T2D. However, there are currently no established methods for providing support to high-risk individuals from different cultural and social backgrounds to help them adopt beneficial lasting lifestyle changes. Instead of just waiting for Iraqi high-risk individuals to develop T2D, this project will implement and assess lifestyle intervention programs aimed at reducing the risk of developing T2D and tailored to individuals with a different social and cultural background.

The study thus seeks to optimize preventive action in health care and aims to facilitate the adoption of permanent changes in lifestyle in high-risk patients, taking account of cultural and social barriers.

Since T2D is associated with a sedentary lifestyle and develops earlier in men than women and an average 10 years earlier in immigrants from the Middle East than in native Swedes, it is crucial to study pathogenic mechanisms triggering T2D development in relation to sex, lifestyle and ethnic background. The results will provide the basis for deciding how health care providers can actively work to prevent T2D and other lifestyle-associated diseases in this high-risk population that has not been studied before.

DETAILED DESCRIPTION:
In this randomized controlled trial, 308 participants (born in Iraq, living in Malmö, Sweden and at high risk of type 2 diabetes) will be allocated to either a culturally adapted intervention or a control group. The intervention will consist of 10 group counseling sessions focusing on diet, physical activity and behavioral change over 6 months, and the offer of exercise sessions. Cultural adaptation includes gender-specific exercise sessions, and counseling by a health coach community member. The control group will receive the information about healthy lifestyle habits provided by the primary health care center. The primary outcome is change in fasting glucose level. Secondary outcomes are changes in body mass index, insulin sensitivity,physical activity, food habits and health-related quality of life. Measurements will be taken at baseline, after 3 and 6 months. Data will be analyzed by the intention-to-treat approach. The cost-effectiveness during the trial period and over the longer term will be assessed by simulation modeling from patient, health care and societal perspectives.

ELIGIBILITY:
Inclusion Criteria:

* (1) 30 to 75 years of age
* (2) individuals in the baseline survey diagnosed with prediabetes. OR BMI ≥ 28 kg/m2 OR waist >=80 cm in females and >=94cm in males.

Exclusion Criteria:

* pregnancy, severe mental illness, diabetes, and/or cognitive impairment, current CVD or history of CVD events. CVD includes stroke, angina or myocardial infarction (MI), percutaneous transluminal coronary angioplasty (PTCA), congestive heart failure (CHF), coronary artery bypass graft surgery (CABG), transient ischemic attack (TIA) and peripheral vascular disease (PVD) or other physical disorders that prevent physical exercise.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Body weight | 4 months
  measured by study nurses
Physical activity | 4 months
  self-reported
Caloric intake | 4 month
  from food records

SECONDARY OUTCOMES:
QALY | 4 month
  The effectiveness will be measured as change in health related quality in life measures as Quality adjusted life years (QALY)
Glycemic changes | 4 month
  fasting glucose, 2-hr glucose
HbA1C | 4 month
Insulin sensitivity and secretion | 4 month
  insulin sensitivity index and disposition index
Blood lipid profile | 4 month
  LDL, HDL, trilycerides
Blood pressure | 4 month
  systolic and diastolic

CONTACTS AND LOCATIONS:
Overall Officials: Louise Bennet, MD,PhD, Principal Investigator — Region Skane
Locations (1):
- Centre for Primary Health Care Research, Region Skåne and Lund University, Malmo, Skåne County, Sweden

REFERENCES:
- [Background] Bennet L, Odeberg H. Resistance to activated protein C, highly prevalent amongst users of oral contraceptives with venous thromboembolism. J Intern Med. 1998 Jul;244(1):27-32. doi: 10.1046/j.1365-2796.1998.00310.x. PMID 9698021
- [Background] Bennet L, Berglund J. Reinfection with Lyme borreliosis: a retrospective follow-up study in southern Sweden. Scand J Infect Dis. 2002;34(3):183-6. doi: 10.1080/00365540110080070. PMID 12030390
- [Background] Bennet L, Danell S, Berglund J. Clinical outcome of erythema migrans after treatment with phenoxymethyl penicillin. Scand J Infect Dis. 2003;35(2):129-31. doi: 10.1080/0036554021000027009. PMID 12693565
- [Background] Bennet L, Halling A, Berglund J. Increased incidence of Lyme borreliosis in southern Sweden following mild winters and during warm, humid summers. Eur J Clin Microbiol Infect Dis. 2006 Jul;25(7):426-32. doi: 10.1007/s10096-006-0167-2. PMID 16810531
- [Background] Bennet L, Fraenkel CJ, Garpmo U, Halling A, Ingman M, Ornstein K, Stjernberg L, Berglund J. Clinical appearance of erythema migrans caused by Borrelia afzelii and Borrelia garinii--effect of the patient's sex. Wien Klin Wochenschr. 2006 Sep;118(17-18):531-7. doi: 10.1007/s00508-006-0659-1. PMID 17009065
- [Background] Jarefors S, Bennet L, You E, Forsberg P, Ekerfelt C, Berglund J, Ernerudh J. Lyme borreliosis reinfection: might it be explained by a gender difference in immune response? Immunology. 2006 Jun;118(2):224-32. doi: 10.1111/j.1365-2567.2006.02360.x. PMID 16771857
- [Background] Bennet L, Stiernstedt S, Berglund J, Hagberg L, Karlsson M, Olsson I, Ornstein K. [Penicillin V is the first choice in the treatment of erythema migrans]. Lakartidningen. 2006 May 3-9;103(18):1454; author reply 1455. No abstract available. Swedish. PMID 16729462
- [Background] Bennet L, Stjernberg L, Berglund J. Effect of gender on clinical and epidemiologic features of Lyme borreliosis. Vector Borne Zoonotic Dis. 2007 Spring;7(1):34-41. doi: 10.1089/vbz.2006.0533. PMID 17417955
- [Background] Ingelsson E, Bennet L, Ridderstrale M, Soderstrom M, Rastam L, Lindblad U. The PPARGC1A Gly482Ser polymorphism is associated with left ventricular diastolic dysfunction in men. BMC Cardiovasc Disord. 2008 Dec 11;8:37. doi: 10.1186/1471-2261-8-37. PMID 19077249
- [Background] Leao TS, Sundquist J, Frank G, Johansson LM, Johansson SE, Sundquist K. Incidence of schizophrenia or other psychoses in first- and second-generation immigrants: a national cohort study. J Nerv Ment Dis. 2006 Jan;194(1):27-33. doi: 10.1097/01.nmd.0000195312.81334.81. PMID 16462552
- [Background] Wang X, Sundquist J, Zoller B, Memon AA, Palmer K, Sundquist K, Bennet L. Determination of 14 circulating microRNAs in Swedes and Iraqis with and without diabetes mellitus type 2. PLoS One. 2014 Jan 30;9(1):e86792. doi: 10.1371/journal.pone.0086792. eCollection 2014. PMID 24497980
- [Background] Arvidsson D, Lindblad U, Sundquist J, Sundquist K, Groop L, Bennet L. Vigorous physical activity may be important for the insulin sensitivity in immigrants from the Middle East and native Swedes. J Phys Act Health. 2015 Feb;12(2):273-81. doi: 10.1123/jpah.2013-0222. Epub 2014 May 6. PMID 24809593
- [Background] Bennet L, Groop L, Lindblad U, Agardh CD, Franks PW. Ethnicity is an independent risk indicator when estimating diabetes risk with FINDRISC scores: a cross sectional study comparing immigrants from the Middle East and native Swedes. Prim Care Diabetes. 2014 Oct;8(3):231-8. doi: 10.1016/j.pcd.2014.01.002. Epub 2014 Jan 25. PMID 24472421
- [Derived] Olaya-Contreras P, Balcker-Lundgren K, Siddiqui F, Bennet L. Perceptions, experiences and barriers to lifestyle modifications in first-generation Middle Eastern immigrants to Sweden: a qualitative study. BMJ Open. 2019 Oct 19;9(10):e028076. doi: 10.1136/bmjopen-2018-028076. PMID 31630098
- [Derived] Siddiqui F, Lindblad U, Nilsson PM, Bennet L. Effects of a randomized, culturally adapted, lifestyle intervention on mental health among Middle-Eastern immigrants. Eur J Public Health. 2019 Oct 1;29(5):888-894. doi: 10.1093/eurpub/ckz020. PMID 30809646
- [Derived] Siddiqui F, Koivula RW, Kurbasic A, Lindblad U, Nilsson PM, Bennet L. Physical Activity in a Randomized Culturally Adapted Lifestyle Intervention. Am J Prev Med. 2018 Aug;55(2):187-196. doi: 10.1016/j.amepre.2018.04.016. PMID 30031454
- [Derived] Saha S, Leijon M, Gerdtham U, Sundquist K, Sundquist J, Arvidsson D, Bennet L. A culturally adapted lifestyle intervention addressing a Middle Eastern immigrant population at risk of diabetes, the MEDIM (impact of Migration and Ethnicity on Diabetes In Malmo): study protocol for a randomized controlled trial. Trials. 2013 Sep 3;14:279. doi: 10.1186/1745-6215-14-279. PMID 24006857